CLINICAL TRIAL: NCT00990314
Title: An Open-label Extension of BPS-MR-PAH-203 in Pulmonary Arterial Hypertension (PAH) Patients
Brief Title: Extension of BPS-MR-PAH-203 in Pulmonary Arterial Hypertension (PAH) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPS-MR-PAH-204
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B.I.D (Experimental): Beraprost Sodium Modified Release Tablet, 60mcg, B.I.D (twice a day dosing)
  Interventions: Drug: Beraprost Sodium Modified Release
- Q.I.D (Experimental): Beraprost Sodium Modified Release Tablet, 60mcg, q.i.d (four times a day dosing)
  Interventions: Drug: Beraprost Sodium Modified Release

INTERVENTIONS:
Drug: Beraprost Sodium Modified Release
  Other Names: BPS-MR Tablets, 60mcg; Beraprost Sodium Modified Release Tablet, 60mcg

SUMMARY:
This is an open-label study for patients who participated in the BPS-MR-PAH-203 study and have volunteered to continue treatment for PAH with Beraprost Sodium Modified Release (BPS-MR) tablets.

DETAILED DESCRIPTION:
Eligible patients who participated in BPS-MR-PAH-203 and who elect to continue receiving study drug in an open-label extension.Each patient will return to the clinic following enrollment in the study at 3, 6, and 12 months, and annually thereafter for assessment. Patients will be called by study personnel to assess adverse events and concomitant medications at Month 9, and at 3 month intervals following the annual visit.

At the End of Study visit, patients discontinuing study drug will be down-titrated off of BPS-MR at the discretion of the Investigator, at a maximum decrement of one tablet (60µg) b.i.d. per day and a minimum decrement of one tablet (60µg) b.i.d. per week. Likewise, patients who withdraw early from the study will be down-titrated off of BPS-MR in the same manner. Upon completion of down-titration, patients will return to the clinic for a final Closeout visit.

Currently enrolled patients may be invited to participate in an optional four times daily (QID) dosing substudy of BPS-MR with total daily dose of BPS-MR achieved previously in the main study. Patients will return to the clinic for baseline visit, week 12, and then will follow the visit schedule provided to them in BPS-MR-PAH-204 main study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who remained on study drug and completed all assessments during the Treatment Phase of Study BPS MR PAH 203 are eligible for this study.
* Women of child-bearing potential (defined as less than 1 year post-menopausal or not surgically sterile) must be using an acceptable method of birth control or practicing abstinence. If sexually active, female patients must use a double barrier method of birth control, such as a condom and spermicidal.

Exclusion Criteria:

* Patients who discontinued study drug during the previous study (BPS MR PAH 203) for any reason (e.g. treatment related adverse events) are not eligible for entry into this study.
* Patients who are pregnant or lactating are excluded from participation in the open-label extension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Smart, Study Director — Study Sponsor
Locations (17):
- United States (6):
  - Harbor-UCLA Medical Center, Torrance, California
  - Midwest Heart Foundation - Advocate Medical Group, Oakbrook Terrace, Illinois
  - Beth Israel Medical Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
- Belgium (2):
  - Universite Libre de Bruxelles, Brussels
  - Catholic University of Leuven, Leuven
- General Teaching Hospital, Prague, Czechia
- Germany (4):
  - Klinikum der Universitat zu Koln, Cologne
  - Medizinische Klinik und Poliklinik, Dresden
  - Abt Innere Medizin III, Medizinische Universitatsklinik, Heidelberg
  - Universitatsklinik Leipzig Abteilung Pulmologie, Leipzig
- Mater Misericordiae University Hospital Ltd., Dublin, Ireland
- Romania (3):
  - Institutul de Urgenta pentru Boli, Bucharest
  - Institutul National de Pneumologie, Bucharest
  - Institutul de Boli Cardiovasculare, Lasi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A Protocol Amendment was to include an optional arm investigating Beraprost Sodium Modified Release Tablets administered four times daily (QID), however, no participants were enrolled into this arm.
Groups:
- Beraprost Sodium: Beraprost Sodium Modified Release Tablet, 60 micrograms(mcg), twice a day dosing
Period: Overall Study
Arm/Group | Beraprost Sodium
Started | 31
Completed | 19
Not Completed | 12
Not completed — Death | 2
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 3
Not completed — Non-Compliance | 1
Not completed — Physician Decision | 3
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Six-Minute Walk Distance [Mean (Standard Deviation); unit: meters] — Area used for the Six Minute Walk Test (6MWT) was pre-measured at 30 meters in length. Rest periods were allowed if patient could no longer continue. If patient needed to rest, he/she could stand or sit and then begin again when rested but the clock continued to run. At the end of 6 minutes, the tester called "stop" while stopping the watch and then measured the distance walked. For purposes of the 6MWT, if patient was assessed at Baseline using oxygen therapy, all future 6MWT were conducted in the same manner. All efficacy results are descriptive; no statistical analysis was conducted. Population: Baseline characteristics were defined as those recorded at the baseline visit of the lead-in study, BPS-MR-PAH-203.
  meters | 360.7 (78.0)
Borg Dyspnea Score [Mean (Standard Deviation); unit: score] — Modified 0-10 category-ratio Borg scale consists of 11-point scale rating the max level of dyspnea experienced during the 6MWT. Scores range from 0 (best condition) and 10 (worst condition) with nonlinear spacing of verbal descriptors of severity corresponding to specific numbers. Participant chose number or verbal descriptor to reflect presumed ratio properties of sensation or symptom intensity. Only participants with both a measurement at baseline and at the given visit are presented. All efficacy results are descriptive; no statistical analysis was conducted. Population: Baseline characteristics were defined as those recorded at the baseline visit of the lead-in study, BPS-MR-PAH-203.
  score | 3.2 (1.97)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least One Treatment-Emergent Adverse Event (TEAE)
Description: A treatment-emergent adverse event (TEAE) is defined as an event not present prior to the initiation of the treatment or any event already present that worsens in either intensity or frequency following exposure to the treatment. AEs occurring more than 3 days after the last day study drug was taken in the study was not included in the statistical analyses or summaries (except for subjects with adverse events leading to study drug withdrawn). Only TEAEs that occurred during the treatment period of the BPS-MR-PAH-204 study were summarized. Any adverse event starting prior to the first dose of study drug was excluded from the summary analyses and only presented in the data listings. All efficacy results are descriptive; no statistical analysis was conducted
Time Frame: Up to 42 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 31
Participants | 27

2. Secondary Outcome: Change in Six-Minute-Walk Distance (6MWD)
Description: Area used for the Six Minute Walk Test (6MWT) was pre-measured at 30 meters in length. Rest periods were allowed if patient could no longer continue. If patient needed to rest, he/she could stand or sit and then begin again when rested but the clock continued to run. At the end of 6 minutes, the tester called "stop" while stopping the watch and then measured the distance walked. For purposes of the 6MWT, if patient was assessed at Baseline using oxygen therapy, all future 6MWT were conducted in the same manner. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline and 42 months
Population: Only participants with both a measurement at Baseline and at the End of Study visit are presented.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 22
meters | 24.09 (81.01)

3. Primary Outcome: Number of Reported Treatment-Emergent Adverse Events
Description: as for outcome 1
Time Frame: Up to 42 months
Measure: Number; unit: TEAEs
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 31
TEAEs | 230

4. Secondary Outcome: Change in Borg Dyspnea Score
Description: The modified 0-10 category-ratio Borg scale consists of an 11-point scale rating the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (for the best condition) and 10 (for the worst condition) with nonlinear spacing of verbal descriptors of severity corresponding to specific numbers. The participant chose the number or the verbal descriptor to reflect presumed ratio properties of sensation or symptom intensity. Baseline was defined as the last non-missing evaluation preceding the first dose of study drug in study BPS-MR-PAH-203. Only participants with both a measurement at baseline and at the given visit are presented. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline and 42 months
Population: Only participants with both a measurement at Baseline and at the End of Study visit are presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 22
scores on a scale | 0.86 (1.89)

5. Secondary Outcome: Number of Participants That Experienced Clinical Worsening
Description: Number of Participants that experienced Clinical Worsening in the opinion of the Investigator. Clinical Worsening was defined as any of these events following the Baseline visit: Death, Transplantation or atrial septostomy, Clinical deterioration as defined by: Hospitalization as a result of PAH symptoms or Initiation of any new PAH specific therapy (e.g. ERA, PDE-5 inhibitor, prostanoid). All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Up to 42 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 31
Participants
  Death | 1
  Hospitalization As A Result of PAH Symptoms | 2
  New PAH Therapies | 4
  Transplantation or atrial septostomy | 0

6. Secondary Outcome: Number of Participants With a Change in WHO Functional Class
Description: Change from Baseline in participant clinical status was recorded according to the World Health Organization (WHO) Functional Class. A change from lower to higher functional class (i.e. 'III to IV' or 'II to III') was considered as a deterioration. A change from higher to lower functional class (i.e. 'III to II' or 'II to I') was considered as an improvement. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline and 42 months
Population: Only participants with both a measurement at Baseline and at the End of Study visit are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 25
Participants
  Improved: Change from Class II to Class I | 2
  Improved: Change from Class III to Class II | 7
  Deteriorated: Change from Class II to Class III | 5
  Deteriorated: Change from Class III to Class IV | 1
  No Change in Class | 10

ADVERSE EVENTS:
Time Frame: From baseline to 30 days after study treatment discontinuation, up to 42 months.
Arm/Group | Beraprost Sodium
All-Cause Mortality (participants affected / at risk) | 2/31
Serious Adverse Events (participants affected / at risk) | 11/31
Other Adverse Events (participants affected / at risk) | 26/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Beraprost Sodium (N=31)
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Worsening pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Edema peripheral (General disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Varicella (Infections and infestations) | 1
Extremity necrosis (Vascular disorders) | 1
Bronchitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Beraprost Sodium (N=31)
Headache (Nervous system disorders) | 10
Nausea (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 5
Fatigue (General disorders) | 5
Flushing (Vascular disorders) | 5
Palpitations (Cardiac disorders) | 4
Upper Respiratory Tract Infection (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 3
Nasopharyngitis (Infections and infestations) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Carbon dioxide decreased (Investigations) | 2
Chest Pain (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 2
Hot flush (Vascular disorders) | 2
Neutrophil count increased (Investigations) | 2
Oedema (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Somnolence (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Tooth abscess (Infections and infestations) | 2
Urine analysis abnormal (Investigations) | 2
Vomiting (Gastrointestinal disorders) | 2
White blood cell count increased (Investigations) | 2
Brain natriuretic peptide increased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days